CLINICAL TRIAL: NCT05410002
Title: A Study on the Effect Diet Has Affecting the Response of Patients Taking N-111 Who Are on a Vegetarian Diet Vs a Non-vegetarian Diet or a Placebo
Brief Title: Diet Effect on Cancer Treatment Outcome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Optimal Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: N-111012422
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Cancer Breast; Cancer Prostate
Keywords: Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized interventional parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active product (N-111) and placebo will be in identical packets with the contents of identical weight, color and texture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Vegetarian N-111 group (Active Comparator): The group will use a vegetarian diet with the active compactor N-111.
  Interventions: Dietary Supplement: Dietary Supplement: N-111
- Non-vegetarian N-111 group. (Active Comparator): The group will use a non-vegetarian diet with the active compactor N-111.
  Interventions: Dietary Supplement: Dietary Supplement: N-111
- Vegetarian placebo group (Placebo Comparator): The group will use a vegetarian diet with a placebo.
  Interventions: Other: Placebo
- Non-vegetarian placebo control group (Placebo Comparator): The group will use a non-vegetarian diet with a placebo.
  Interventions: Other: Placebo
- Vegetarian control group (No Intervention): The group will use a vegetarian diet without the active compactor N-111 or the placebo.
- Non-vegetarian control group (No Intervention): he group will use a non-vegetarian diet without the active compactor N-111 or the placebo.

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: N-111 — Dietary supplement N-111
  Arms: Non-vegetarian N-111 group.; Vegetarian N-111 group
Other: Placebo — Dietary placebo
  Arms: Non-vegetarian placebo control group; Vegetarian placebo group

SUMMARY:
The study will look at the end result of 2 types of diets effect on treatment outcome of cancer patients using N-111.

DETAILED DESCRIPTION:
The study will be evaluated during a double blind, placebo-controlled evaluation of the effect diet has on the response of patients taking N-111 who are on a vegetarian diet vs a non-vegetarian diet or a placebo. This will involve assessing the patients progress or lack thereof over a 3-month period of time as outlined in Outcome Measures section below.

ELIGIBILITY:
Inclusion Criteria:

* A positive diagnosis of breast cancer as determined by Fine Needle Biopsy or open biopsy with associated Cancer Antigen blood markers.
* Prostate cancer as determined by a Transrectal Biopsy with associated Prostate- specific antigen blood work.

Exclusion Criteria:

* •Patients without the positive diagnosis of breast or prostate cancer.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Active Comparator: Vegetarian N-111 group | End of month 3.
  Change in blood levels (CA, CMP, CBC, CEA, Lipids, CRP) from base line to the end of month 3.
Active Comparator: Non-vegetarian N-111 group. | End of month 3.
  Change in blood levels (CA, CMP, CBC, CEA, Lipids, CRP) from base line to the end of month 3.

SECONDARY OUTCOMES:
Placebo Comparator: Vegetarian placebo group | End of month 3.
  Change in blood levels (CA, CMP, CBC, CEA, Lipids, CRP) from base line to the end of month 3.
Placebo Comparator: Non-vegetarian placebo control group | End of month 3.
  Change in blood levels (CA, CMP, CBC, CEA, Lipids, CRP) from base line to the end of month 3.

CONTACTS AND LOCATIONS:
Overall Officials: EA Jeppsen, MD, Study Chair — Optimal Health Research
Locations (3):
- Optimal Health Research, Salt Lake City, Utah, United States
- India (2):
  - KLE Academy of Higher Education & Research, Belagāve, Karnataka
  - Indian Institute of Research, Mumbai

IPD SHARING:
Plan to Share IPD: No